CLINICAL TRIAL: NCT04430010
Title: Multi-level Determinants of Implementation and Sustainment in the Education Sector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20019081; R01MH124439 (NIH)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Evidence Based Programs in Schools
MeSH Terms: interventions — Bestrophins; Artifacts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation (Experimental): Teachers will implement the BEST in CLASS treatment in their classrooms
  Interventions: Behavioral: BEST in CLASS

INTERVENTIONS:
Behavioral: BEST in CLASS — BEST in CLASS is a Tier-2 evidence based program (EBP) that has demonstrated effectiveness at reducing children's Disruptive Behavior Problems (DBPs) and risk for Emotional and Behavioral Disorders (EBDs)

SUMMARY:
The purpose of this study is to learn more about teachers' sustainment of use of core components of BEST in CLASS in a follow-up study.

DETAILED DESCRIPTION:
The goal of this study is to help understand how to successfully implement and sustain evidence based programs (EBP) in the education sector. The study will look at how questions such as what teacher, program, and school characteristics impact sustainment of the EBP BEST in CLASS, what modifications to BEST in CLASS represent a sustained program, and how do teacher, program, and school characteristics influence sustainment of BEST in CLASS.

ELIGIBILITY:
Inclusion Criteria:

Teacher participants

* teach in general education Kindergarten, 1st, 2nd, or 3rd grade
* consent to participate
* proficient in English
* participated as a BEST in CLASS teacher who received coaching in the prior year

Family participants

* proficient in English
* have a school-age child or children
* consent to participate

Children participants

* enrolled in a general Kindergarten, 1st, 2nd or 3rd grade classroom
* proficient in English
* at elevated risk for EBD
* demonstration of externalizing behaviors that interfere with participation in the classroom (e.g., disruption, aggression) as indicated by teacher rating
* parental/guardian consent to participate

Exclusion Criteria:

Teacher participants

* do not teach in general education Kindergarten, 1st, 2nd, or 3rd grades
* were not part of the BEST in CLASS intervention condition in the year prior
* do not consent to participate
* do not speak fluent English
* do not have at least one student that meets the inclusion criteria

Family participants

* do not speak proficient English
* do not provide consent
* do not have elementary aged children will be excluded.

Children participants

* caregivers do not provide permission for participation
* caregiver(s) do not speak proficient English
* are not proficient in English
* do not screen in as demonstrating risk for EBD

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Program Adherence | baseline to 9 months
  Change in the degree to which the teacher adheres to the BEST in CLASS treatment during observations as measure by the TREATMENT INTEGRITY INSTRUMENT FOR ELEMENTARY SETTINGS (TIES) Adherence scale. The TIES-A is an 18 item scale of BEST in CLASS practices. Teachers are rated on the presence (use) of each practice on a scale from 1 (not at all) to 7 (extensively). Scores are summed giving a range of 18 to 126. Higher scores are associated with greater adherence.
Change in Program Competence | baseline to 9 months
  Change in the degree to which the teacher adheres to the BEST in CLASS treatment during observations as measure by the TREATMENT INTEGRITY INSTRUMENT FOR ELEMENTARY SETTINGS (TIES) Competence scale. The TIES-C is an 18 item scale of BEST in CLASS practices. For all practices observed (greated than 1 on the Adherence scale) teachers are rated on the competency of their use of the practice on a scale from 1 (not at all) to 7 (extensively). Scores are summed giving a range of 0 to 126. Higher scores are associated with greater competence.
Change in student disruptive behavior problems | Baseline to 9 months
  Student disruptive behaviors will be measured by the Social Skills Improvement System (SSIS) total problems scale. Higher scores represent more problem behaviors.
Change in student prosocial behavior | Baseline to 9 months
  Student prosocial behaviors will be measured by the Social Skills Improvement System (SSIS) social skills scale. Higher scores represent more prosocial behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Bryce D McLeod, PhD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No